CLINICAL TRIAL: NCT03058302
Title: Study of Effectiveness and Implementation of Different Versions of the CETA Mental Health Intervention Among Internally Displaced Persons (IDPs) and Veterans in Ukraine
Brief Title: Study of Effectiveness and Implementation of a Mental Health Intervention With Conflict-affected Communities in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7293
Record Dates: First submitted 2017-02-13; First posted 2017-02-20 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Depression; PostTraumatic Stress Disorder
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: until the 4th sessions participants receiving CETA and providers will be masked with respect to whether treatment is short or long CETA.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full CETA (Experimental): Full CETA participants will complete 12 CETA sessions. this is the same version of CETA that has been tested in other sites. They will be monitored weekly for clinical purposes (symptoms and safety) during treatment. they will also receive monthly research assessments (research outcomes) for 6 months after baseline assessment and commencement of treatment.
  Interventions: Behavioral: CETA (Common Elements Treatment Approach)
- Brief CETA (Experimental): Brief CETA participants is a new shorter version of CETA that has the same content as Full CETA but provided in fewer sessions. Each participant will complete 5 CETA sessions and will be monitored weekly for clinical purposes (symptoms and safety) during treatment and thereafter monthly for research purposes (research outcomes) for 6 months after baseline assessment and commencement of treatment.
  Interventions: Behavioral: CETA (Common Elements Treatment Approach)
- Wait-Control (No Intervention): Wait-control participants will undergo monthly monitoring after enrollment in the study for research purposes (research outcomes) for 6 months after baseline assessment.

INTERVENTIONS:
Behavioral: CETA (Common Elements Treatment Approach) — The Common Elements Treatment Approach, or CETA, is a transdiagnostic psychotherapy based on cognitive behavioral elements for mood, anxiety and trauma related problems. CETA is based on the fact that most evidence-based mental health treatments (EBTs) consist of similar components. The objective of CETA is to provide a single training in a range of therapy components that are similar across EBTs and to then teach counselors how to design a specific course of treatment for each client based on the client's presenting problems.
  Arms: Brief CETA; Full CETA

SUMMARY:
This project aims to contribute to the development of a community mental health care system while directly serving the conflict affected population in east Ukraine. This project is being supported by USAID's Victims of Torture Fund. In the Spring of 2015, the Johns Hopkins University (JHU) Applied Mental Health Research Group (AMHR) was invited to make a site visit to Ukraine with USAID to make an initial assessment of current mental health problems, service capacities, and treatment need. AMHR and USAID were requested by community-based partners to provide training and support in evidence based trauma treatment for people affected by war and displacement. Extensive conflict within the borders of Ukraine is a new experience for most Ukrainians, and local psychologists and psychotherapists were not prepared for wide-spread need or trained in appropriate methods of treatment for affected populations. JHU and USAID began activities in Ukraine in June 2015 and have identified the counseling intervention, Common Elements Treatment Approach (CETA), as appropriate and relevant for this context. Community providers from the three trial sites (Kyiv, Kharkiv, and Zaporizhia) have been trained in CETA as counselors and local supervisors.

An ongoing training and supervision model (Apprenticeship Model) is being implemented in the three study sites. These three sites contain significant numbers of military veterans (demobilized soldiers from the ongoing conflict) and internally displaced persons (IDPs). Adult IDPs and Veterans from the three study sites will be recruited and screened to identify those with elevated depression and/or posttraumatic stress symptoms and impaired functioning. This study will be conducted as a 3-armed randomized controlled trial. This study will test to see if both the long and a short version of CETA are effective compared to a wait-control condition.

DETAILED DESCRIPTION:
This research team developed the CETA intervention and has evaluated its effectiveness in multiple trials. CETA was developed based on other transdiagnostic interventions that have proven efficacious in the United States and Europe. Briefly, full length CETA includes 12 weekly treatment sessions comprised of cognitive behavioral elements. In the last few years, as more researchers have identified mental health interventions that can successfully reduce the burden of symptoms for clients in low-resource settings, there has been a push to develop intervention models that are more scalable. One of the barriers to scalability may be duration of treatment, as clients may not complete treatment if there are too many sessions, and counselors may be limited in the number of clients they can treat over the course of a year when each client requires more sessions. However, the trade-off of potential reduction in treatment efficacy has not been evaluated for shortened- versus standard-length treatment models of efficacious interventions. This study will begin to address this by testing to see if both the long and a short version of CETA are effective compared to wait-control condition. Community providers from the three trial sites (Kyiv, Kharkiv, and Zaporizhia) have begun ongoing training in CETA as counselors and local supervisors.

This study will be conducted as a 3-armed randomized controlled trial. Adult IDPs, Ukrainian military veterans, and their family members in 3 Ukrainian cities, Kyiv, Kharkiv, and Zaporizhia, will be recruited on a rolling basis and screened to identify those with elevated depression and/or posttraumatic stress (PTS) symptoms and impaired functioning using a locally validated assessment instrument. Local non-governmental organizations (NGOs) and existing service providers have been provided with a locally validated short clinical assessment instrument (developed during a previous phase of the current research). As part of regular services, these organizations will use this instrument to assess their clientele for need for specific clinical services. If the assessment suggests that the person is in need of services and the person agrees to seek help they will then refer them to the study's monitoring and evaluation (M&E) staff who will meet with each potential participant and conduct a repeat screening to ensure trial eligibility. Those who meet the eligibility criteria on this second screen will be consented for the study. All eligible and consented adults will be randomly allocated to either a wait-list control condition, the Brief CETA model, or the Full CETA model. After randomization, those allocated to either CETA arm will be referred to one of the local counselors or supervisors, all of whom are trained in both versions of CETA (Brief and Full). for purposes of blinding those allocated to a CETA arm (and their counselors) will not be aware of whether they are receiving the full CETA (12 sessions) or the short CETA (5 sessions). This information will be revealed to the provider and client after the 4 session, so that they can plan either to end treatment at the 5th session or continue. All study participants in all 3 arms will be assessed on a monthly basis for 6 months post-baseline. After completion of their participation in the trial those assigned to the wait-control condition will be able to receive CETA services.

At the 1st monthly data collection point post treatment completion, study participants in the short CETA and long CETA intervention arms will also be interviewed using a Client Dissemination and Implementation Research (D&I) instrument that explores aspects of program implementation from the client perspective. In addition, the first 30 participants (total N=60) to complete both versions of CETA will also be asked to provide a qualitative interview upon completion of their treatment exploring unexpected effects of the program, both positive and negative. Data from these D&I interviews will be used to improve the program. Data from the qualitative interview will also be used generate additional locally important items to add to the study impact assessment instruments. This expanded version of the instrument will be completed by later study participants.

CETA providers (counselors and supervisors) will be interviewed after 6 months of providing CETA services using both a Provider Dissemination and Implementation (D&I) instrument and a qualitative interview. The purpose of the provider D&I instrument is similar to that for the clients, but from the provider perspective (i.e., to identify aspects of program implementation that should be changed in order to improve the program). The purpose of the qualitative interview is the same as the D&I instrument but to identify unknown factors affecting implementation that are not referred to in the instrument. important local information from the latter will not be added to the D&I instrument but will be included in reports as qualitative data only.

Primary Aim:

1. To determine the effectiveness of 2 versions of CETA (brief: 5 sessions; full: 12 sessions) in comparison with a wait-list control condition for reducing the severity of depression and posttraumatic stress symptoms and improving daily functioning experienced by IDPs and veterans in Ukraine.

   Secondary Aims:
2. To explore the effectiveness of each version of CETA in comparison with a wait-list control condition for reducing anxiety symptom severity and reducing substance abuse (alcohol and drug) among IDPs and veterans in Ukraine.
3. To explore provider and participant level factors affecting CETA implementation.

ELIGIBILITY:
Inclusion Criteria:

* Ukrainian adults (age 18 or older) who are either Internally Displaced Persons (IDPs) or military veterans of the conflict is East Ukraine, and their adult family members.
* A score of 7 or above on the locally validated depression scale AND a score of 4 or above on the locally validated function scale
* A score of 9 or above on the locally validated PTS scale AND a score of 4 or above on the locally validated function scale
* Living in or around the 3 study sites for the duration of the study (at least 6 months) and able to regularly attend at least one of the locations where CETA is available for duration of treatment.

Exclusion Criteria:

* Our definition of "veteran" excludes people who identify as veterans but are still active (i.e., active duty) in the Ukrainian military.
* Active thoughts and plans of suicidality or symptoms of psychosis requiring immediate referral to professional psychiatric services.
* Factors identified at baseline that preclude full participation, including: unstable and severe medical, psychiatric or drug use problem that currently necessitates inpatient treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-01; Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Change in Mental health symptom levels from baseline (monthly for all groups) | Monthly for 6 months
  Change in Symptoms of depression and posttraumatic stress from baselines, measured monthly for all groups for 6 months post baseline
Change in Impaired functioning levels (monthly for all groups) | 6 months post-baseline
  Change in Impaired functioning levels from baseline, measured at the 6 month follow-up for all groups.

SECONDARY OUTCOMES:
Change in Mental health symptom levels from baseline (Monthly for all groups) | Monthly for 6 months
  Change in Symptoms of anxiety and alcohol use from baseline, measured monthly for all groups for 6 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolton, MBBS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Laura Murray, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Ukraine (3):
  - National University of Kyiv Mohyla Academy, Kharkiv
  - National University of Kyiv Mohyla Academy, Kyiv
  - National University of Kyiv Mohyla Academy, Zaporozh’ye

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared with other collaborators and researchers. Data that is not de-identified will never be shared.

REFERENCES:
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Background] McHugh RK, Murray HW, Barlow DH. Balancing fidelity and adaptation in the dissemination of empirically-supported treatments: The promise of transdiagnostic interventions. Behav Res Ther. 2009 Nov;47(11):946-53. doi: 10.1016/j.brat.2009.07.005. Epub 2009 Jul 29. PMID 19643395
- [Background] Murray LK, Dorsey S, Haroz E, Lee C, Alsiary MM, Haydary A, Weiss WM, Bolton P. A Common Elements Treatment Approach for Adult Mental Health Problems in Low- and Middle-Income Countries. Cogn Behav Pract. 2014 May;21(2):111-123. doi: 10.1016/j.cbpra.2013.06.005. PMID 25620867
- [Derived] Murray LK, Haroz EE, Doty B, Singh NS, Bogdanov S, Bass J, Dorsey S, Bolton P. Testing the effectiveness and implementation of a brief version of the Common Elements Treatment Approach (CETA) in Ukraine: a study protocol for a randomized controlled trial. Trials. 2018 Aug 3;19(1):418. doi: 10.1186/s13063-018-2752-y. PMID 30075806